CLINICAL TRIAL: NCT01746758
Title: Establishing a Community Referral System to Improve Uptake of Adolescent Sexual Reproductive Health Services in Mwanza, Tanzania
Brief Title: Mobile Phone Text Messaging Referral
Acronym: SMS4Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Ministry of Health and Social Welfare, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11.94RS
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-05

CONDITIONS: HIV; Sexually Transmitted Infections; Contraception; Pregnancy
Keywords: Reproductive health, mHealth, Cluster randomised trial
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS text messaging referral (Experimental): The text messaging system has been designed to use codes of reproductive health conditions and their treatments. Text messages are sent by drug stores and received at the dispensaries, forwarded by a bespoke software called Snapshot, which captures data online from any computer anywhere by use of a login for confidentiality.
  Interventions: Behavioral: SMS text messaging referral
- Comparison arm (No Intervention): No intervention will be implemented in intervention arm. Data on reproductive health conditions and treatments and data on referrals from drug stores in this arm will be obtained directly from ministry of health registers filled and filed at the dispensary and health centres, plus a tailor-made form which is filled by the dispensary and health centre clinicians whenever they receive a patient in the eligible categories.

INTERVENTIONS:
Behavioral: SMS text messaging referral — The text messaging system has been designed to use codes of reproductive health conditions and their treatments. Text messages are sent by drug stores and received at the dispensaries, forwarded by a bespoke software called Snapshot, which captures data online from any computer anywhere by use of a login for confidentiality.
  Arms: SMS text messaging referral

SUMMARY:
The study hypothesis is that managed referral of patients at community level (from drug stores) increases uptake of reproductive health (RH) services at dispensary and health centre levels.

The intervention is currently being implemented in 2 districts (Magu and Sengerema) in Mwanza Region on the northwest shore of Lake Victoria. It is nested within the IntHEC Community Randomised Trial which aims to evaluate the impact of a complex RH intervention on the uptake and integration of reproductive health services in 2 Regions in Tanzania (Mwanza and Iringa) and Niger (Say and Aguie) respectively. 18 wards per region were stratified according to geographical and economic criteria and randomly assigned to intervention or comparison wards. The SMS intervention is being implemented in 9 intervention wards in Mwanza Region only. 9 wards are followed for comparison.

DETAILED DESCRIPTION:
The SMS intervention was developed in 2 phases: (i) stakeholder consultation and (ii) technical design. Twenty-three consultation meetings were held with 78 drug store owners and attendants, 45 dispensary and health centre clinical officers and nurses, and 148 adolescents in communities. These stakeholders prioritised key deficiencies in existing RH provision and preferred strategies to address them. Detailed methods and results of these consultations are presented elsewhere (Consultation Paper in preparation). In brief government health facilities wanted an intervention that allows dispensaries and health centres to take charge of STI treatment and provide skilled service for other RH needs. Drug stores wanted an intervention that recognises and integrates their contribution to the health system, while adolescents wanted an intervention that promotes accessibility, confidentiality and trust of service providers. Through subsequent meetings, an SMS intervention strategy was identified because all clinical officers and drug store attendants demonstrated use mobile phones on a day-to-day basis.

The intervention design prioritised patients' ease of access to service: when a patient comes to a drug store to buy medicines for a RH related problem that may require a prescription drug, the drug store explains the referral system. If the patient accepts, the drug store sends a text message with the patient details to a toll-free number connected to a web-system. The system processes and forwards the patient details including a password to a dispensary matched with the referrer drug store. At the same time, that password is sent back to the referrer drug store so that it can be passed on to the patient. While at dispensary, patients with a password are received, matched with details received in text messages, and given fast track RH service, after which the dispensary sends a text message to the toll-free number confirming the completeness of patient treatment. This intervention is implemented in all 9 intervention wards in Mwanza. No intervention is implemented in the 9 comparison wards.

ELIGIBILITY:
Inclusion Criteria:

Only patients attending services at the drug store. Only patients seeking reproductive health care services. Only resident in study wards.

Exclusion Criteria:

Patients non-residence in study wards. Patients seeking non-reproductive health care services.

The primary and secondary outcomes will be measured in people aged 15-19 (our definition of adolescent), but the intervention accepts all age-groups during implementation.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Increase the number of patients receiving reproductive health services at dispensary and health centre level after referral from a drug store. | 12 months
  This will be measured by comparing data of referred patients by text message in intervention wards with patients' data from comparison wards - comparing the number of referrals from drug stores in both arms.

SECONDARY OUTCOMES:
Referred number of patients attending HIV, STI, pregnancy prevention (including numbers of condoms, VCT, and post-abortion care) and treatment | 12 months
  Obtained from data on the text messaging system and from comparison communities
Referred number of patients attending other contraceptives (the pill, intra-uterine devices, injection, female condom and sterilisation where available) | 12 months
  Obtained from data on the text messaging system and from comparison communities
Referred number of patients testing HIV positive (where there is a testing service) | 12 months
  Obtained from data on the text messaging system and from comparison communities
Referred number of patients diagnosed with STIs (syndromic diagnosis) | 12 months
  Obtained from data on the text messaging system and from comparison communities
Prevalence of HIV and STIs in the data from study areas | 12 months
  Obtained from data on the text messaging system and from comparison communities

CONTACTS AND LOCATIONS:
Overall Officials: John N Dusabe, MSc BSc, Principal Investigator — Liverpool School of Tropical Medicine; Angela IN Obasi, MSc PhD MRCP, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- National Institute for Medical Research Tanzania, Mwanza, Tanzania